CLINICAL TRIAL: NCT05738135
Title: Effect of Intravenous Aminophylline on Hemodynamics and Recovery of Patients Undergoing Functional Endoscopic Sinus Surgery Under Dexmedetomidine Hypotensive Anesthesia: A Randomized Controlled Study
Brief Title: Aminophylline on Recovery in Functional Endoscopic Sinus Surgery Under Dexmedetomidine Hypotensive Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, Lecturer of Anesthesiology, Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36264PR58/1/23
Record Dates: First submitted 2023-02-11; First posted 2023-02-21 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-03

CONDITIONS: Aminophylline; Dexmedetomidine; Functional Endoscopic Sinus Surgery
Keywords: Aminophylline; Dexmedetomidine; Hemodynamics; Recovery; Functional Endoscopic Sinus Surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aminophylline group (Experimental): Patients will receive 4 mg/kg aminophylline diluted in 50 ml normal saline over 30 minutes.
  Interventions: Drug: Aminophylline group
- Control group (Placebo Comparator): Patients will receive 50 ml normal saline over 30 minutes.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Aminophylline group — Patients will receive 4 mg/kg aminophylline diluted in 50 ml normal saline over 30 minutes.
  Arms: Aminophylline group
Drug: normal saline — Patients will receive 50 ml normal saline over 30 minutes.
  Arms: Control group

SUMMARY:
This study will be conducted to evaluate the effect of intravenous aminophylline on hemodynamics and recovery of patients receiving dexmedetomidine infusion during functional endoscopic sinus surgery.

DETAILED DESCRIPTION:
Aminophylline is a nonselective adenosine receptor antagonist used for the treatment of asthma and chronic obstructive pulmonary disease. It has been used to antagonize the effects of anaesthetic and analgesic agents

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 50 years, have American society of anesthesiology (ASA) physical status I - II and scheduled for elective FESS under general anesthesia and receiving dexmedetomidine infusion for controlled hypotension during surgery.

Exclusion Criteria:

1. Patients with central nervous system diseases, cardiovascular diseases, hypertension, arrhythmias, cerebrovascular diseases, convulsions, renal impairment or hepatic dysfunction.
2. Pregnancy or lactation.
3. Patients with a history of allergy to aminophylline.
4. Patients with recurrent sinus surgery, hypertension.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Time to extubation | Two hours after discontinuation of anesthetics
  Extubation time, defined as the interval between the discontinuation of anesthetics to safe tracheal extubation.

SECONDARY OUTCOMES:
Intraoperative heart rate | Intraoperative period
  Heart rate will be recorded preoperatively (baseline), after loading dose of dexmedetomidine, after intubation, every 5 minutes during the study drug infusion, then every 15 minutes until end of surgery.
Intraoperative mean arterial blood pressure | Intraoperative period
  Mean arterial blood pressure will be recorded preoperatively (baseline), after loading dose of dexmedetomidine, after intubation, every 5 minutes during the study drug infusion, then every 15 minutes until end of surgery.
Postoperative sedation score | 60 minutes after tracheal extubation
  Postoperative sedation will be evaluated using the Ramsay sedation score as:
  1 = anxious, agitated, or restless 2= cooperative, oriented, and tranquil 3= responsive to commands 4= a sleep, but with brisk response to light, glabella tap, or loud auditory stimulus 5= a sleep, sluggish response to glabella tap, or auditory stimulus 6= a sleep, no response 6 is the highest sedation level Sedation score: will be measured at 15, 30, and 60 minutes after tracheal extubation.
Time to discharge from post anesthesia care unit | Two hours after tracheal extubation.
  Time needed to achieve modified Aldrete Score ≥9 will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding after 6 mon from publication
Supporting Information: Study Protocol, SAP
Time Frame: after 6 mon from publication
Access Criteria: The data will be available upon reasonable request from the corresponding